CLINICAL TRIAL: NCT00347139
Title: Multi-centre, Randomised, Double-blind, Placebo-controlled, Four-way Incomplete Block Crossover Study, to Examine Efficacy, Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single and Repeat Administration of Three Inhaled Doses (25, 100 and 400 mcg Once Daily) of GW642444
Brief Title: Repeat Doses Of A New Medication (GW642444) In Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B2C106093
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Tolerability; Pharmacodynamics; Safety; Pharmacokinetics; GW642444; Asthmatic patients; Efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- GW642444 (Experimental)
  Interventions: Drug: GW642444 (25, 100 & 400 mcg/day)
- Salmeterol (Active Comparator)
  Interventions: Drug: Salmeterol 50mcg

INTERVENTIONS:
Drug: GW642444 (25, 100 & 400 mcg/day) — 25, 100 and 400mcg/dose
  Arms: GW642444
Drug: Salmeterol 50mcg — Salmeterol 50mcg
  Arms: Salmeterol

SUMMARY:
In order to obtain information on a wider range of doses of GW642444 (a possible new medication to treat asthma) than has been previously examined in asthmatic patients, this current study will be conducted at doses of 25 100 and 400 mcg of GW642444 and will be compared with salmeterol (50 mcg twice daily). This study will be conducted in a similar manner to a study that has already been completed (study number B2C101762) which examined repeat doses of 50, 100 and 200 mcg of GW642444. The data obtained will compliment the data from study B2C101762 and will provide confidence (or not) that the desired bronchodilation can be achieved and maintained without undesirable side effects.

ELIGIBILITY:
Inclusion criteria:

* Subjects with a documented history of persistent asthma.
* Current non-smokers.
* Clinically stable persistent asthma FEV1 between 60 and 90% of predicted values.
* Inhaled corticosteroid therapy at a total daily dose between 200-500mcg of fluticasone or equivalent.

Exclusion criteria:

* Subjects with significant past or present disease which which may affect their safety.
* Upper or lower respiratory tract infection within 4 weeks of screening.
* History of life threatening asthma, or asthma requiring treatment with oral corticosteroids within 3 months of study.
* Patients taking doses of inhaled corticosteroid >500mcg/day and patients who have changed therapy within 8 weeks of the study.
* Patients weighing less than 50kg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-05-23 (Actual); Primary Completion 2007-01-10 (Actual); Study Completion 2007-01-10 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline (pre-dose on Day 1) in the mean of 23 and 24 hour (h) visit (pre-bronchodilator and pre-dose) trough FEV1 after repeat dosing over 14 days | From Baseline (pre-dose on Day 1) and up to 14 days
  The forced expiratory volume in one second (FEV1) is the amount of air exhaled in one second after an forceful inspiration. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline was defined as the value recorded pre-dose (before dosing) on Day 1. Least square mean change along with standard error has been presented.

SECONDARY OUTCOMES:
Mean change from Baseline (pre-dose on Day 1) in weighted mean clinic FEV1 on Day 1 and Day 14 | From Baseline (pre-dose on Day 1) and at 0-2 h, 0-4, and 0-24 h Days 1 and 14
  The forced expiratory volume in one second is the amount of air exhaled in one second after an forceful inspiration. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline was the pre-dose value recorded on Day 1. Weighted means have been presented as least square means. Analysis performed using mixed effect ANCOVA with fixed effects covariates of baseline FEV1, center, sex, age, treatment period, treatment and the mean of the participants Baseline values. Participant was fitted as a random coefficient.
Mean change from Baseline (pre-dose on Day 1) in morning (AM) Peak expiratory flow rate (PEFR) from electronic flow meter over Days 2-15 | Baseline (pre-dose on Day 1) and up to 15 days
  The forced expiratory volume in one second is the amount of air exhaled in one second after an forceful inspiration. Change from Baseline is the value at indicated time point minus the Baseline value. AM PEFR values were measured by electronic flow meter. PEFR is maximum speed of expiration of participant as measured by the device and AM PEFR was calculated in each morning, over period. Analysis performed using mixed effect ANCOVA with fixed effects covariates of Baseline AM PEFR, center, sex, age, treatment period, treatment and the mean of the participants Baseline values. Participant was fitted as a random coefficient. Least square mean change along with standard error has been presented.
Mean change from Baseline (pre-dose on Day 1) in the evening (PM) PEFR from electronic flow meter over Days 1-14 | Baseline (pre-dose on Day 1) and up to 14 days
  The forced expiratory volume in one second is the amount of air exhaled in one second after an forceful inspiration. Change from Baseline is the value at indicated time point minus the Baseline value. PM PEFR values were measured by electronic flow meter. PEFR is maximum speed of expiration of participant as measured by the device and PM PEFR was calculated in each evening over period. Analysis performed using mixed effect ANCOVA with fixed effects covariates of Baseline PM PEFR, center, sex, age, treatment period, treatment and the mean of the participants Baseline values. Participant was fitted as a random coefficient. Least square mean change along with standard error has been presented.
Mean change from Baseline (pre-dose on Day 1) in AM FEV1 from electronic flow meter over Days 2-15 | Baseline (pre-dose on Day 1), Day 2, and Day 15
  The forced expiratory volume in one second is the amount of air exhaled in one second after an forceful inspiration. Change from Baseline is the value at indicated time point minus the Baseline value. AM FEV1 values were measured by electronic flow meter and was measured in the morning over period. Analysis performed using mixed effect ANCOVA with fixed effects covariates of baseline AM FEV1, center, sex, age, treatment period, treatment and the mean of the participants Baseline values. Participant was fitted as a random coefficient. Least square mean change along with standard error has been presented.
Mean change from Baseline (pre-dose on Day 1) in PM FEV1 from electronic flow meter over 14 days | Baseline (pre-dose on Day 1) and up to Day 14
  The forced expiratory volume in one second is the amount of air exhaled in one second after an forceful inspiration. Change from Baseline is the value at indicated time point minus the Baseline value. PM FEV1 values were measured by electronic flow meter and was measured in the evening over period. Analysis performed using mixed effect ANCOVA with fixed effects covariates of Baseline PM FEV1, center, sex, age, treatment period, treatment and the mean of the participants Baseline values. Participant was fitted as a random coefficient. Least square mean change along with standard error has been presented.
Change in AM PEFR from Pre-AM Dose to Post-AM Dose at Day1, 7, and 14 | Day 1, 7, and 14
  The forced expiratory volume in one second is the amount of air exhaled in one second after an forceful inspiration. Change in post-AM PEFR is the value at indicated time point minus the pre-AM PEFR value. AM PEFR values were measured by electronic flow meter. PEFR is maximum speed of expiration of participant as measured by the device and AM PEFR was calculated in each morning, over period.
Change in PM PEFR from Pre-PM Dose to Post-PM Dose at Day1, 7, and 14 | Day 1, 7, and 14
  The forced expiratory volume in one second is the amount of air exhaled in one second after an forceful inspiration. Change in post-PM PEFR is the value at indicated time point minus the pre-PM PEFR value. PM PEFR values were measured by electronic flow meter. PEFR is maximum speed of expiration of participant as measured by the device and PM PEFR was calculated in each morning, over period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Germany (2):
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
- GSK Investigational Site, Wellington, New Zealand
- GSK Investigational Site, Moscow, Russia
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: B2C106093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C106093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2C106093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C106093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C106093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C106093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2C106093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register